CLINICAL TRIAL: NCT04225806
Title: Investigation of Femoropopliteal In Situ Valve Formation With the InterVene System (INFINITE-US)
Acronym: INFINITE-US
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project suspended by Sponsor
Sponsor: Intervene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN004
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Venous Insufficiency (CVI); Deep Vein Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Investigational (Experimental): Subjects will be treated with the investigational device and followed per protocol.
  Interventions: Device: BlueLeaf® Endovenous Valve Formation System (BlueLeaf System)

INTERVENTIONS:
Device: BlueLeaf® Endovenous Valve Formation System (BlueLeaf System) — The BlueLeaf System is a single-use, disposable device designed to modify the vein wall to form one or more functional autogenous valves to improve the hemodynamics of the deep venous system treated.

SUMMARY:
Prospective, non-randomized, multicenter pre-market early feasibility study (EFS) to evaluate subjects treated with the BlueLeaf System for the treatment of symptomatic chronic venous insufficiency (CVI) of the lower extremity

DETAILED DESCRIPTION:
The purpose of this early feasibility study is to provide information on the BlueLeaf System for the formation of one or more autogenous vein valves constructed from the vein wall of the femoral and/or popliteal vein, in subjects with CVI and who meet the specified eligibility criteria. In particular, the safety and technical feasibility of the procedure will be validated in patients in the United States, including the procedural steps, operator technique, and subject characteristics. The study will assess the safety and effectiveness of the study device acutely and through 5 years.

ELIGIBILITY:
Key Inclusion Criteria

* Failed at least 6 months of conservative therapy at some point during the course of their CVI management (symptoms not adequately resolved or patient non-compliant/unable to tolerate)
* Deep system venous reflux characterized by >1 second reflux time in two vein segments (vein segments defined as: proximal femoral, distal femoral, and popliteal), as assessed by duplex ultrasound (DUS) with patient in the standing position
* Presence of at least two potential target sites within a target vessel as assessed preliminarily by DUS, with a target site being defined as a segment within the femoral or popliteal vein that is:

  7mm to 11mm in luminal diameter and at least 3cm long and absent features that, in the Investigator's opinion, would preclude formation of a monocuspid valve (at any orientation).
* In the Investigator's opinion, the subject is a good candidate for treatment with the BlueLeaf System based on their symptoms, quality of life, anatomy, and the likelihood of benefit from continued conservative therapy

Key Exclusion Criteria:

* Untreated significant superficial venous incompetence which, in the opinion of the Investigator, may be the primary source of existing symptoms
* Acute deep venous thrombosis (DVT) within 1 year of consent
* Deep venous intervention (includes stenting) in the target limb or outflow vessels within 3 months of consent
* Flow-limiting venous outflow obstruction central to the intended target sites, defined by a common femoral vein duplex exam found to have a continuous waveform without respiratory variation
* Contraindications to all protocol specified anticoagulation options
* Known and uncontrolled hypercoagulopathy (i.e. hypercoagulopathy that cannot be adequately managed/controlled with medication)
* Women on long-term oral contraceptives
* Non-ambulatory patients
* Significant peripheral arterial disease with an ankle-brachial index of < 0.70 or with incompressible vessels
* New York Heart Association Class III or IV heart failure
* Patients with a history of right heart failure occurring as a consequence of, for example, biventricular failure, intrinsic pulmonary disease, chronic thromboembolic pulmonary hypertension, and other etiologies that result in elevated right-sided pressures.
* Active systemic infection
* Invasive surgical procedure within the last 3 months that in the Investigator's opinion would interfere with the study procedure or results
* Chronic renal insufficiency with creatinine level of ≥ 2mg/dL
* Hemoglobin level < 9.0 mg/dL
* Platelet count < 50,000 or > 1,000,000/mm3
* Total white blood cell count < 3,000/mm3
* Subject is enrolled in another clinical study that, in the opinion of the Investigator, may conflict with this study or compromise study results
* Comorbidity risks or other concerns which, in the opinion of the Investigator, either limits longevity or likelihood of complying with the protocol and its prescribed follow up (e.g. recent cancer or stroke); or precludes patient from being transitioned to open surgery if complication requiring surgical intervention occurs during the procedure (such as severe vein laceration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Elkins, Study Director — Intervene, Inc.
Locations (5):
- United States (5):
  - The Vascular Experts, Darien, Connecticut
  - NYU Langone Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Sentara Vascular Specialists, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational
Started | 15
Completed | 0 (Trial was terminated prior to the last protocol-mandated follow-up at 5 years post-procedure.)
Not Completed | 15
Not completed — Trial termination | 15

BASELINE CHARACTERISTICS:
Arm/Group | Investigational
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Revised Venous Clinical Severity Score (rVCSS) [Median (Standard Deviation); unit: score on a scale] | 14.4 (4.2)
Deep Venous Thrombosis (DVT) [Count of Participants; unit: Participants]
  Right | 5
  Left | 3
  Bilateral | 1
  None | 6
Diabetes [Count of Participants; unit: Participants]
  Type 1 | 0
  Type 2 | 3
  None | 12
Smoker [Count of Participants; unit: Participants]
  Current | 2
  Former | 6
  Never | 7
Chronic Kidney Disease [Count of Participants; unit: Participants]
  Yes | 2
  No | 13
History of Stroke [Count of Participants; unit: Participants]
  Yes | 0
  No | 15
History of Malignancy [Count of Participants; unit: Participants]
  Yes, active | 0
  Yes, inactive | 1
  No | 14
History of Peripheral Artery Disease (PAD) [Count of Participants; unit: Participants]
  Yes, active | 1
  Yes, inactive | 0
  No | 14
History of Hypercoagulable Syndrome [Count of Participants; unit: Participants]
  Yes, active | 2
  Yes, inactive | 0
  No | 13
History of Coronary Artery Disease [Count of Participants; unit: Participants]
  Yes | 1
  No | 14
History of Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants]
  Yes | 1
  No | 14
History of Pulmonary Embolism [Count of Participants; unit: Participants]
  Yes | 3
  No | 12
History of Chronic Venous Insufficiency (CVI) [Count of Participants; unit: Participants]
  Yes | 15
  No | 0
Prior Superficial Vein Treatment [Number; unit: procedures]
  None | 7
  Surgical stripping/ligation | 4
  Foam sclerotherapy | 3
  Endovenous ablation/closure | 7
History of Congestive Heart Failure (CHF) [Count of Participants; unit: Participants]
  Yes | 1
  No | 14
Prior Deep Venous System or Outflow Vessel Intervention [Number; unit: participants]
  Yes | 7
  No | 8
Prior Fem-pop Balloon Angioplasty [Number; unit: procedures]
  Right | 2
  Left | 0
  Bilateral | 1
Prior Thrombectomy [Number; unit: procedures]
  Right | 0
  Left | 0
  Bilateral | 0
Prior Venous Stenting [Number; unit: procedures]
  Right | 2
  Left | 2
  Bilateral | 0
Prior Venous Valve Reconstruction Surgery [Number; unit: procedures]
  Right | 0
  Left | 0
  Bilateral | 0
Prior Inferior Vena Cava (IVC) Filter Placement [Count of Participants; unit: Participants]
  Yes, filter still present | 2
  Yes, filter not present | 1
  No | 12
History of Corona Virus Disease 2019 (COVID-19) [Count of Participants; unit: Participants]
  Previous | 1
  Current | 0
  None | 12
  Unknown | 2
Clinical-Etiology-Anatomy-Pathophysiology (CEAP) Classification [Count of Participants; unit: Participants]
  C3 - edema | 0
  C4 - changes in skin and subcutaneous tissue secondary to chronic venous disease | 0
  C5 - healed | 7
  C6 - active venous ulcer | 3
  C6r - recurrent active venous ulcer | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: The Number of Subjects Experiencing a Major Adverse Event (MAE), Composed of the Following
Description: * Symptomatic pulmonary embolism
  * DVT anywhere in the deep venous system of the treatment limb
  * Occlusive valve pocket thrombus (VPT)
  * Non-occlusive stenosis in the target vessel (including due to scarring, inflammation, VPT, etc.) leading to persistent worsening of symptoms attributable to venous flow obstruction, or requiring post-procedural surgical or endovascular re-intervention
  * Device or procedure-related venous or arterial injury in the treated limb (such as Arteriovenous Fistula (AVF's), bleeding, pseudo aneurysm) leading to worsening of symptoms that require post-procedural surgical or endovascular re-intervention or requiring transfusion of more than 2 units of blood. (Note: Peri-procedural stiches placed to assist with closure of the access site will not be characterized as a primary safety failure.)
  * Device or procedure-related death
Time Frame: 30-day post-procedure
Population: All subjects that were treated with the investigational device
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational
Number analyzed (Participants) | 15
Participants | 0

2. Primary Outcome: Change in Revised Venous Clinical Severity Score (rVCSS) From Baseline
Description: Assessment of changes in the rVCSS; the score is a composite based on a rating score of none (0), mild (1), moderate (2) and severe (3) for symptoms and clinical signs, the number of active ulcers (0, 1, 2, >/=3), duration of ulcers (<3 months, >3 months but <1 year, not healed for >1 year), active ulcer size (diameter <2cm, diameter 2-6cm, and diameter >6cm), and use of compression therapy (not used (0), intermittent use of stockings (1), wears stockings most days (2), and full compliance (3)). A higher VCSS would indicate a worse outcome.
Time Frame: Baseline, 30-days, 12-weeks, 210-days and 365-days post-procedure
Population: Only available data is reported and therefore, the number analyzed may differ across the timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational
Number analyzed (Participants) | 15
score on a scale
  Baseline Score | 14.1 (4.2)
  30-day Score | 13.5 (5.4)
  Change from Baseline - 30-day | -0.4 (5.5)
  12-week Score: number analyzed (Participants) | 14
  12-week Score | 12.6 (4.8)
  Change from Baseline - 12-week: number analyzed (Participants) | 14
  Change from Baseline - 12-week | -1.4 (5.4)
  210-day Score: number analyzed (Participants) | 12
  210-day Score | 11.3 (5.3)
  Change from Baseline - 210-day: number analyzed (Participants) | 12
  Change from Baseline - 210-day | -2.4 (4.3)
  365-day Score: number analyzed (Participants) | 14
  365-day Score | 11.5 (4.8)
  Change from Baseline - 365-day: number analyzed (Participants) | 14
  Change from Baseline - 365-day | -2.3 (4.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Investigational
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=15)
Infection (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) — event occurred due to a fall resulting in a large left hip hematoma
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cellulitis (Injury, poisoning and procedural complications) | 1 (1) — cellulitis of right lower extremity
Hypotension (Cardiac disorders) | 1 (1)
Bleeding varicosity (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=15)
Chest pressure (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal bruising (Musculoskeletal and connective tissue disorders) | 2 (2)
Achilles tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Allergic reaction with blistering on skin (Injury, poisoning and procedural complications) | 1 (1)
Groin complication (Injury, poisoning and procedural complications) | 1 (1) — event is a consequence of the angiography procedure
Animal Bite (Injury, poisoning and procedural complications) | 1 (1)
Arthritis flare (Immune system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain post-procedure (Injury, poisoning and procedural complications) | 1 (1) — attributed to the positioning of the participant during the procedure
Contusion of right thigh (Injury, poisoning and procedural complications) | 1 (1)
Epistaxis (General disorders) | 1 (1)
Essential hypertension (Cardiac disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Flu (Infections and infestations) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
Indeterminate thrombus (Vascular disorders) | 1 (1)
Infection at enoxaparin injection site (Infections and infestations) | 1 (1)
Injection site reactions (Injury, poisoning and procedural complications) | 1 (1)
Left Lateral ankle venous ulcer infection (Infections and infestations) | 1 (1)
Leg cramps index leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bleeding at lovenox injection site (General disorders) | 1 (1)
New venous ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in chest and arms (bilateral) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Post procedure bleeding at access site (Injury, poisoning and procedural complications) | 1 (1)
Posterior left knee soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Recurrent left ankle ulcer infection (Infections and infestations) | 1 (1)
Renal stones with hydroureteronephrosis (Renal and urinary disorders) | 1 (1)
Right ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right thumb cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Right toe cellulitis (Infections and infestations) | 1 (1)
Sore throat (General disorders) | 1 (1)
ST depression (Cardiac disorders) | 1 (1)
Tinnitus Left ear (Ear and labyrinth disorders) | 1 (1)
Valve Pocket Thrombus (VPT) (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1)
Venous ulcer infection (Infections and infestations) | 4 (8)
Worsening osteoarthritis left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening ulceration relating to infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial was terminated early by Sponsor, and therefore, analysis of data is limited to available information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT04225806/Prot_SAP_000.pdf